CLINICAL TRIAL: NCT03809455
Title: Effectiveness and Tolerance of Fentanyl Citrate in Painful Pain Induced During Diagnostic or Therapeutic Examinations in Cancer Patients
Acronym: FARADI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled by Sponsor.
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UC-0106/1607 SdS 02 FARADI
Record Dates: First submitted 2018-10-11; First posted 2019-01-18 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough Pain
MeSH Terms: conditions — Breakthrough Pain | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: A phase II, prospective, multicentre, single-blinded, randomised study (when fentanyl citrate is used outside of its marketing authorisation) Patients will be enrolled in an observational cohort when the fentanyl citrate is used according to its marketing authorisation.
  The study will randomise patients (2:1; FAR Arm: Placebo Arm)
  Stratified by:
  * Centre
  * Type of examination: diagnostic (PET-CT scan or SPECT-CT scan) versus therapeutic (radiotherapy, tomotherapy, or dosimetric scanner)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAR Arm (Experimental)
  Interventions: Drug: Fentanyl citrate
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl citrate — Fentanyl citrate arm (FAR Arm): one intake of fentanyl citrate 100 µg (intranasal or buccal).
  Placebo Arm: one intake of placebo (intranasal or buccal) The administration route will be left to the discretion of the investigator taking into account the patient's profile (capable of maintaining the sublingual tablet without swallowing, absence of nasal discharge…), and/or the patient's choice.
  Medication Commercial name Formulation Administration route Dose Fentanyl citrate Pecfent® Nasal spray Intranasal 100 µg Fentanyl citrate Abstral® Sublingual tablet Buccal 100 µg For the cohort the choice of treatment by FAR is at the centres discretion, according to standard of practice.
  Treatment duration: 1 day
  Arms: FAR Arm
Drug: Placebo — one intake of placebo (intranasal or buccal)
  Arms: Placebo Arm

SUMMARY:
A phase II, prospective, multicentre, single-blinded, randomised study (when fentanyl citrate is used outside of its marketing authorisation) Patients will be enrolled in an observational cohort when the fentanyl citrate is used according to its marketing authorisation.

DETAILED DESCRIPTION:
Primary objective (phase II trial):

Evaluate the efficacy of an administration of fentanyl citrate to alleviate breakthrough pain caused by positional requirements of a diagnostic or therapeutic intervention/examination in cancer patients who do not meet the prescription criteria for fentanyl citrate's marketing authorisation, as follows:

* Patients having received less than 60 mg of slow-release/extended-release morphine.
* Patients having received slow-release/extended-release morphine for less than 7 days.
* Patients who have not received any opioid treatment.

Primary objective (cohort):

Evaluate the efficacy of an administration of fentanyl citrate to alleviate breakthrough pain caused by positional requirements of a diagnostic or therapeutic intervention/examination in cancer patients when used within the marketing authorisation, as follows:

* Patients having at least 60 mg of slow-release/extended-release morphine.
* Patients having received slow-release/extended-release morphine for at least 7 days.
* Patients who have already received an opioid treatment (at least equivalent to 60 mg /day of oral morphine) for chronic cancer-related pain for at least 7 days.

Secondary objectives (phase II and cohort):

* Evaluate the tolerance of the administration of fentanyl citrate when used to alleviate breakthrough pain caused by positional requirements of a diagnostic or therapeutic intervention/examination in cancer patients.
* Evaluate the efficacy of fentanyl citrate for reducing pain.
* Evaluate the efficacy of fentanyl citrate for reducing anxiety.
* Evaluate the percentage of relief and patients' satisfaction related to the administration of fentanyl citrate.

Secondary objectives (phase II only):

• Describe the reasons why the diagnostic or therapeutic intervention/examination failed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients in follow up or being treated for cancer.
3. Patients with cancer-related pain (area of pain located near primary tumor or metastatic lesions).
4. Patients:

   1. not having received any opioid treatment (opioid naïve).
   2. or, treated for less than 7 days by a slow-releasing/extend-release opioid treatment; and/or by less than 60 mg per day of oral morphine, or less than 30 mg/day of oral oxycodone, or less than 8 mg/day of oral hydromorphone, or less than 25 µg/h of transdermal fentanyl.
5. Patients need to have at least one of the following interventions, lasting between 25 and 45 minutes during which they will be request to not move:

   1. Radiotherapy session*, including tomography (patients hospitalized or treated as outpatients).
   2. Dosimetric scanner (hospitalized patients).
   3. Positron-emission tomography** (PET): PET-computed tomography [CT] scan and single photon emission computed tomography [SPECT]-CT scan (hospitalized patients).
6. Public health insurance coverage.

(*) A patient who has numerous radiotherapy sessions can only be included once; (**) with acquisition phase in a prostrate or decubitus dorsal position and strictly immobile in one of the cameras (PET or SPECT).

Inclusion criteria (cohort):

As for the inclusion criteria for the phase II study, with the following modifications:

4. Patients treated with a slow-releasing/extended-release opioid for:

1. more than 7 days.
2. and with at least 60 mg per day of oral morphine, or at least 30 mg/day of oral oxycodone, or at least 8 mg/day of oral hydromorphone, or at least 25 µg/h of transdermal fentanyl.

   5. Patients who believes that they are cannot assume a prostrate or decubitus dorsal position for a diagnostic or therapeutic examination/intervention due to the pain they will experienced in this position,

   Or

   Patients experience breakthrough pain (numerical pain scale 5), in a region corresponding to the localization of the metastatic lesions or the primary tumor, when they assume a prostrate/decubitus dorsal position,

   Or

   Patients who have breakthrough pain (numerical pain scale 5) in a region corresponding to the localization of the metastatic lesions or the primary tumor that prevents the completion of a diagnostic or therapeutic examination/intervention.

   6. Public health insurance coverage.

   Exclusion Criteria:
   1. Patients with contraindication for the administration of fentanyl citrate: severe respiratory depression or a severe obstructive pulmonary disease.
   2. Patients who have already participated in this study.
   3. Patients with a history of alcoholism or substance/drug dependence.
   4. Patients with an intravenous or subcutaneous opioid patient-controlled analgesic (PCA) pump.
   5. Patients unable to communicate or understand instructions in French.
   6. Patients deprived of their liberty or under protective custody or guardianship, or unable to provide their consent for study participation.
   7. Patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Successful diagnostic or therapeutic examination | 1 hours after randomization
  A patient will be considered a success if the planned immobilization period is completed.